

Statistical data was expressed as standard deviation (SD) for continuously changing data and as percentile (%) for median and categorical variables. Wilcoxon rank-sum test or t-test were used based on parametric or non-parametric data for continuous variables to compare the differences between survivors and non-survivors. The survival rate was shown with the Kaplan-Meier estimator curve. Univariate and multivariate logistic regression models were used to investigate risk factors associated with death in intensive care.